CLINICAL TRIAL: NCT00362141
Title: Safety and Tolerability of Add-on Levetiracetam in Status Epilepticus
Brief Title: Safety and Tolerability Study of Levetiracetam to Treat Patients With Status Epilepticus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Center Haaglanden (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-013; METC 06-013
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2007-04-02 (Estimated); Status verified 2007-03

CONDITIONS: Status Epilepticus
Keywords: levetiracetam; status; epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levetiracetam (add-on)

SUMMARY:
The purpose of this study is to determine whether levetiracetam is safe and well tolerated by patients while suffering a status epilepticus. Levetiracetam is added to the standard treatment of patients with this disease.

DETAILED DESCRIPTION:
Status epilepticus (SE) is a disorder with high mortality and morbidity. There are strong indications that ongoing seizure activity substantially reduces the chances on a good outcome. This implies that optimal treatment of SE should start as soon as possible. Unfortunately, treatment options are limited and often based on little evidence. Besides, current treatment options are hampered by serious side-effects like respiratory depression and impaired consciousness. Therefore, the advent of new and effective anti-epileptic drugs (AEDs) is of great potential interest for the treatment of SE. Presently, the newer AEDs are mainly used in later stages of SE at a time when the disease is often more difficult to control. The characteristics of one of these recently introduced anticonvulsants i.e. levetiracetam seems to provide a number of fortunate properties for application as first-line treatment of SE. The complicating side-effects of "classical" AEDs, like a decrease in cardiorespiratory function or in level of consciousness are hardly present. Besides, levetiracetam may lower the need for benzodiazepines, reducing chances on respiratory depression by benzodiazepines at higher doses. Due to a remarkable synergism with first-line administered benzodiazepines, levetiracetam may therefore reduce the need for intubation or ICU treatment. Besides, it may enhance the immediate cessation of seizures, prolong the anti-seizure activity of benzodiazepines and provide neuroprotective properties. The sustained efficacy of levetiracetam would suggest that long term sequelae secondary to neurological damage, may also be reduced. Levetiracetam IV has recently been shown to be safe in healthy volunteers, and becomes available for iv application in clinical practice, early 2006. To date, there are hardly any data available on its applicability in medical emergencies like SE. We propose as a first step the executing of a phase II study on tolerability and safety of intravenous levetiracetam in patients with SE. Current first-line treatment of SE consists of standardized administration of benzodiazepines. For the study we propose to apply this regimen together with the iv administration of levetiracetam as add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years of age
* All types of SE, diagnosed by the medical examiner according to the predefined definition. Absence SE has to be confirmed by EEG.
* Woman: 18-50 years of age of whom is known, from anamnesis or hetero-anamnesis (first line relative), that she is not pregnant.

Exclusion Criteria:

* Woman < 50 years of age, without information on pregnancy
* Known pregnancy
* Known allergy for levetiracetam
* Daily dose levetiracetam of more than 2000mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-10; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
o Uneventful intravenous (iv) administration of study medication
o Toxicity profile on iv administration, including:
§ Irritation on injection site
§ Hypotension, defined as systolic blood pressure below 90 mm Hg recorded within 24 hours of the dose
§ Cardiac arrest (diagnosed clinically) or bradyarrhythmias including heart block, documented on an electrocardiogram
§ Respiratory depression, defined as the occurrence of apnea or need for intubation
§ Allergic reactions, like skin rash
§ Other side-effects

SECONDARY OUTCOMES:
Pharmacokinetic parameters of levetiracetam and clonazepam in patients with SE

CONTACTS AND LOCATIONS:
Overall Officials: Charles Vecht, MD, PhD, Principal Investigator — Medical Centre Haaglanden
Locations (1):
- Medical Centre Haaglanden, The Hague, South Holland, Netherlands

REFERENCES:
- See also: CCMO — http://www.ccmo-online.nl